CLINICAL TRIAL: NCT00000414
Title: Patient Education Strategies for Better Outcomes in Rheumatoid Arthritis (RA) and Osteoarthritis (OA)
Brief Title: Patient Education in Rheumatoid Arthritis and Osteoarthritis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: National Institute of Arthritis and Musculoskeletal and Skin Diseases (NIAMS) (NIH)
Responsible Party: Principal Investigator, Kate Lorig, professor, Stanford University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P01 AR43584 Substudy 004; P01AR043584 (NIH)
Record Dates: First submitted 1999-11-03; First posted 1999-11-04 (Estimated); Last update posted 2013-06-21 (Estimated); Status verified 2004-11

CONDITIONS: Rheumatoid Arthritis; Osteoarthritis
Keywords: Rheumatoid arthritis (RA); Osteoarthritis (OA); Arthritis education; Health care service evaluation; Outcomes research; Arthritis Self-Management Program (ASMP); Self-Managed Arthritis Relief Therapy (SMART) Program
MeSH Terms: conditions — Arthritis, Rheumatoid; Osteoarthritis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arthritis Self-Management Program (Experimental): small group self-management program
  Interventions: Behavioral: Arthritis Self-Management Program
- SMART Program (Experimental): Self-Managed Arthritis Relief Therapy: mailed self management material
  Interventions: Behavioral: SMART Program

INTERVENTIONS:
Behavioral: Arthritis Self-Management Program
  Arms: Arthritis Self-Management Program
Behavioral: SMART Program
  Other Names: Self-Managed Arthritis Relief Therapy (SMART)
  Arms: SMART Program

SUMMARY:
This project will evaluate the effectiveness and general usefulness of two arthritis patient education programs. The first, the Arthritis Self-Management Program, is a 6-week, community-based program taught in small groups by peer leaders. The second, the Self-Managed Arthritis Relief Therapy (SMART) Program, is a computer-driven program delivered through the mail. Participants in this project are people with rheumatoid arthritis or osteoarthritis who are taking part in the larger long-term studies being conducted by ARAMIS (the Arthritis, Rheumatism and Aging Medical Information System).

DETAILED DESCRIPTION:
In a changing health care environment, the role of patients in managing their arthritis is increasingly important. Patient education is the primary means for teaching patients how to fulfill this role successfully. The goal of self-management health education is not merely to provide information but also to change patient attitudes and behavior so that patient outcomes are improved. These programs represent a new treatment for arthritis.

This project will evaluate the relative effect on health status and cost-effectiveness of two arthritis patient education programs that use different delivery systems. The Arthritis Self-Management Program (ASMP) uses a small group, multi-class format. It is taught by trained lay leaders and has been evaluated for effectiveness and widely disseminated. The Self-Managed Arthritis Relief Therapy (SMART) Program is a computer-driven, individualized, mail-delivered intervention. Results of a pilot study suggest that it is effective in improving health status and reducing health care use.

The project will also evaluate how generalizable the SMART program is and its effectiveness for patients with different diagnoses (OA and RA). It will also determine the attributes of patients who choose and do not choose to participate in patient education programs as well as the attributes of those who complete and do not complete the ASMP and SMART programs.

Through use of the ARAMIS data collection system, the project allows us to describe the differences between people who volunteer to receive patient education and those who refuse patient education. This project is directed at improving patient outcomes in both RA and OA through wide availability of a low-cost, mail-delivered arthritis self-management program that is the next generation in arthritis health education.

ELIGIBILITY:
Inclusion Criteria:

* Physician diagnosis of OA or RA
* Participation in the ARAMIS longitudinal study

Exclusion Criteria:

* Age under 18

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1200 (Actual)
Dates: Start 1996-07; Primary Completion 2001-04 (Actual); Study Completion 2001-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kate R. Lorig, DrPH, Principal Investigator — Stanford University
Locations (5):
- United States (4):
  - Stanford University, Palo Alto, California
  - Wichita Arthritis Center, Wichita, Kansas
  - University of Pittsburgh, Pittsburgh, Pennsylvania
  - Vanderbilt University, Nashville, Tennessee
- University of Saskatoon, Edmonton, Alberta, Canada

REFERENCES:
- [Background] Lorig KR, Ritter PL, Laurent DD, Fries JF. Long-term randomized controlled trials of tailored-print and small-group arthritis self-management interventions. Med Care. 2004 Apr;42(4):346-54. doi: 10.1097/01.mlr.0000118709.74348.65. PMID 15076811